CLINICAL TRIAL: NCT03027011
Title: Effect of Remote Ischemic Preconditioning on Brain Injury in Carotid Endarterectomy
Brief Title: Remote Ischemic Preconditioning on Brain Injury in Carotid Endarterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XYFY-2017-005
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Brain Injuries; Remote Ischemic Preconditioning
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Preconditioning(RIPC) (Active Comparator): RIPC will be induced during anesthesia by 3 cycles of 5-min upper limb ischemia and 5-min reperfusion using a blood-pressure cuff inflated to a pressure 200mmHg
  Interventions: Procedure: Remote Ischemic Preconditioning
- Control (Placebo Comparator): Control group without remote ischemic preconditioning
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — RIPC will be induced during anesthesia by 3 cycles of 5-min upper limb ischemia and 5-min reperfusion using a blood-pressure cuff inflated to a pressure 200mmHg
  Other Names: RIPC
  Arms: Remote Ischemic Preconditioning(RIPC)
Procedure: Control — Control group without remote ischemic preconditioning
  Arms: Control

SUMMARY:
This is a randomized controlled trial designed to test an intervention (Remote ischemic preconditioning) in patients undergoing carotid endarterectomy (CEA).Remote ischemic preconditioning(RIPC) with transient upper limb ischemia/reperfusion is a novel, simple, cost-free,non-pharmacological and non-invasive strategy.The purpose of this study is to evaluate the effects of Remote Ischaemic Preconditioning on perioperative ischaemic injury in patients undergoing carotid endarterectomy compared to control intervention.The outcomes of interest include neurocognitive function,clinical outcomes,and biomarkers of brain injury.

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIPC) protocol will be induced during anesthesia by 3 cycles of 5-min upper limb ischemia and 5-min reperfusion using a blood pressure cuff inflated to a pressure 200mmHg

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing carotid endarterectomy
* Patients aged 55 years to 80 years

Exclusion Criteria:

* Inability to give informed consent
* Known Deep venous thrombosis (DVT) in arm
* Pre-existing lymphedema or axillary node dissection both arms
* Arteriovenous fistula or graft in both arms
* Left ventricular ejection fraction less than 50%
* Diagnosis of dementia, intellectual disability, or mental illness including depression, anxiety, or schizophrenia

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
S100-beta biomarker | 48 hours post surgery
  tested by ELISA

SECONDARY OUTCOMES:
Short - term cognitive function | 1 day before surgery and 1 week post surgery
  Short - term cognitive function will be tested by mini-mental state examination
Neuron specific enolase (NSE) biomarker | 48 hours post surgery
  tested by ELISA
Sleep quality | 1 week post surgery
  Sleep quality will be test by medical outcomes study sleep scale

CONTACTS AND LOCATIONS:
Overall Officials: Chen Xiuxia, MD, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will be available when this trial is finished and the article have been published

REFERENCES:
- [Result] Naylor AR. What is the current status of angioplasty vs endarterectomy in patients with asymptomatic carotid artery disease? J Cardiovasc Surg (Torino). 2007 Apr;48(2):161-80. PMID 17410063
- [Result] Naylor AR. Where next after SPACE and EVA-3S: 'the good, the bad and the ugly!'. Eur J Vasc Endovasc Surg. 2007 Jan;33(1):44-7. doi: 10.1016/j.ejvs.2006.11.002. Epub 2006 Nov 28. PMID 17126572
- [Result] Brevoord D, Kranke P, Kuijpers M, Weber N, Hollmann M, Preckel B. Remote ischemic conditioning to protect against ischemia-reperfusion injury: a systematic review and meta-analysis. PLoS One. 2012;7(7):e42179. doi: 10.1371/journal.pone.0042179. Epub 2012 Jul 31. PMID 22860077
- [Result] Sanderson TH, Reynolds CA, Kumar R, Przyklenk K, Huttemann M. Molecular mechanisms of ischemia-reperfusion injury in brain: pivotal role of the mitochondrial membrane potential in reactive oxygen species generation. Mol Neurobiol. 2013 Feb;47(1):9-23. doi: 10.1007/s12035-012-8344-z. Epub 2012 Sep 26. PMID 23011809
- [Result] Pundik S, Xu K, Sundararajan S. Reperfusion brain injury: focus on cellular bioenergetics. Neurology. 2012 Sep 25;79(13 Suppl 1):S44-51. doi: 10.1212/WNL.0b013e3182695a14. PMID 23008411
- [Result] Bhuiyan MI, Kim YJ. Mechanisms and prospects of ischemic tolerance induced by cerebral preconditioning. Int Neurourol J. 2010 Dec;14(4):203-12. doi: 10.5213/inj.2010.14.4.203. Epub 2010 Dec 31. PMID 21253330
- [Result] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170
- [Result] Przyklenk K, Bauer B, Ovize M, Kloner RA, Whittaker P. Regional ischemic 'preconditioning' protects remote virgin myocardium from subsequent sustained coronary occlusion. Circulation. 1993 Mar;87(3):893-9. doi: 10.1161/01.cir.87.3.893. PMID 7680290
- [Result] Nandagopal K, Dawson TM, Dawson VL. Critical role for nitric oxide signaling in cardiac and neuronal ischemic preconditioning and tolerance. J Pharmacol Exp Ther. 2001 May;297(2):474-8. PMID 11303032
- [Result] Kitagawa K, Matsumoto M, Tagaya M, Hata R, Ueda H, Niinobe M, Handa N, Fukunaga R, Kimura K, Mikoshiba K, et al. 'Ischemic tolerance' phenomenon found in the brain. Brain Res. 1990 Sep 24;528(1):21-4. doi: 10.1016/0006-8993(90)90189-i. PMID 2245337
- [Result] Ederle J, Featherstone RL, Brown MM. Percutaneous transluminal angioplasty and stenting for carotid artery stenosis. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD000515. doi: 10.1002/14651858.CD000515.pub3. PMID 17943745
- [Result] Lim SY, Yellon DM, Hausenloy DJ. The neural and humoral pathways in remote limb ischemic preconditioning. Basic Res Cardiol. 2010 Sep;105(5):651-5. doi: 10.1007/s00395-010-0099-y. Epub 2010 May 7. PMID 20449597
- [Result] Manchurov V, Ryazankina N, Khmara T, Skrypnik D, Reztsov R, Vasilieva E, Shpektor A. Remote ischemic preconditioning and endothelial function in patients with acute myocardial infarction and primary PCI. Am J Med. 2014 Jul;127(7):670-3. doi: 10.1016/j.amjmed.2014.02.012. Epub 2014 Feb 21. PMID 24565591
- [Result] Olguner C, Koca U, Kar A, Karci A, Islekel H, Canyilmaz M, Mavioglu O, Kizildag S, Unlu G, Elar Z. Ischemic preconditioning attenuates the lipid peroxidation and remote lung injury in the rat model of unilateral lower limb ischemia reperfusion. Acta Anaesthesiol Scand. 2006 Feb;50(2):150-5. doi: 10.1111/j.1399-6576.2006.00938.x. PMID 16430534
- [Result] Xia Z, Herijgers P, Nishida T, Ozaki S, Wouters P, Flameng W. Remote preconditioning lessens the deterioration of pulmonary function after repeated coronary artery occlusion and reperfusion in sheep. Can J Anaesth. 2003 May;50(5):481-8. doi: 10.1007/BF03021061. English, French. PMID 12734158
- [Result] Jiang HW, Chen C, Hao LJ. [Protective effect of limb ischemic preconditioning against liver ischemia/reperfusion injury in the rat]. Zhongguo Ying Yong Sheng Li Xue Za Zhi. 2010 Nov;26(4):502-4. Chinese. PMID 21329001
- [Result] Cao L, Yuan G, Wang Y, Chang Y, Xu J, Zou D, Wei L. [Limb ischemic preconditioning reduces rabbit hepatic ischemia-reperfusion injury through inhibition the phosphorylation of proteins in the MAPK signal pathway in the late phase]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2012 Jun;37(6):591-7. doi: 10.3969/j.issn.1672-7347.2012.06.009. Chinese. PMID 22772420
- [Result] Sun XC, Li WB, Li QJ, Zhang M, Xian XH, Qi J, Jin RL, Li SQ. Limb ischemic preconditioning induces brain ischemic tolerance via p38 MAPK. Brain Res. 2006 Apr 21;1084(1):165-74. doi: 10.1016/j.brainres.2006.02.041. Epub 2006 Apr 21. PMID 16631139
- [Result] Rehni AK, Shri R, Singh M. Remote ischaemic preconditioning and prevention of cerebral injury. Indian J Exp Biol. 2007 Mar;45(3):247-52. PMID 17373368
- [Result] Rehni AK, Singh N, Jaggi AS. Possible involvement of insulin, endogenous opioids and calcitonin gene-related peptide in remote ischaemic preconditioning of the brain. Yakugaku Zasshi. 2007 Jun;127(6):1013-20. doi: 10.1248/yakushi.127.1013. PMID 17541253
- [Result] Vlasov TD, Korzhevskii DE, Poliakova EA. [Ischemic adaptation of the rat brain as a method for protection of endothelium from ischemic reperfusion injury]. Ross Fiziol Zh Im I M Sechenova. 2004 Jan;90(1):40-8. Russian. PMID 15143491
- [Result] Hahn CD, Manlhiot C, Schmidt MR, Nielsen TT, Redington AN. Remote ischemic per-conditioning: a novel therapy for acute stroke? Stroke. 2011 Oct;42(10):2960-2. doi: 10.1161/STROKEAHA.111.622340. Epub 2011 Aug 11. PMID 21836089
- [Result] Malhotra S, Naggar I, Stewart M, Rosenbaum DM. Neurogenic pathway mediated remote preconditioning protects the brain from transient focal ischemic injury. Brain Res. 2011 Apr 22;1386:184-90. doi: 10.1016/j.brainres.2011.02.032. Epub 2011 Feb 19. PMID 21338588
- [Result] Hougaard KD, Hjort N, Zeidler D, Sorensen L, Norgaard A, Hansen TM, von Weitzel-Mudersbach P, Simonsen CZ, Damgaard D, Gottrup H, Svendsen K, Rasmussen PV, Ribe LR, Mikkelsen IK, Nagenthiraja K, Cho TH, Redington AN, Botker HE, Ostergaard L, Mouridsen K, Andersen G. Remote ischemic perconditioning as an adjunct therapy to thrombolysis in patients with acute ischemic stroke: a randomized trial. Stroke. 2014 Jan;45(1):159-67. doi: 10.1161/STROKEAHA.113.001346. Epub 2013 Nov 7. PMID 24203849
- [Result] Tulu S, Mulino M, Pinggera D, Luger M, Wurtinger P, Grams A, Bodner T, Beer R, Helbok R, Matteucci-Gothe R, Unterhofer C, Gizewski E, Schmutzhard E, Thome C, Ortler M. Remote ischemic preconditioning in the prevention of ischemic brain damage during intracranial aneurysm treatment (RIPAT): study protocol for a randomized controlled trial. Trials. 2015 Dec 29;16:594. doi: 10.1186/s13063-015-1102-6. PMID 26714784
- [Result] Walsh SR, Nouraei SA, Tang TY, Sadat U, Carpenter RH, Gaunt ME. Remote ischemic preconditioning for cerebral and cardiac protection during carotid endarterectomy: results from a pilot randomized clinical trial. Vasc Endovascular Surg. 2010 Aug;44(6):434-9. doi: 10.1177/1538574410369709. Epub 2010 May 18. PMID 20484064